CLINICAL TRIAL: NCT04391673
Title: Analysis of Illness Perceptions Affecting the Outcome of Vestibular Rehabilitation
Brief Title: Factors Affecting Outcome of Vestibular Rehabilitation
Status: Withdrawn | Type: Observational
Why Stopped: Chief Investigator Moved Hospitals Before the Trial Began. Was discontinued.
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 269318
Record Dates: First submitted 2020-02-05; First posted 2020-05-18 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Chronic Dizziness; Vestibular Disease
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dizzy group: Patients attending the dizziness and balance exercise programme at Guy's Hospital, London. Patients data will be included if they complete at least 4 sessions.
  Interventions: Behavioral: Vestibular rehabilitation

INTERVENTIONS:
Behavioral: Vestibular rehabilitation — Vestibular rehabilitation (treatment as usual).

SUMMARY:
This is an observational longitudinal study to investigate if negative illness perceptions predict less improvement in dizziness handicap following vestibular rehabilitation. Consecutive patients (n=260) who enter the vestibular rehabilitation programme at Guy's Hospital, London will be included. Questionnaires will be conducted immediately before, and after their final treatment. The main outcome will be the Dizziness Handicap Inventory after rehabilitation.

DETAILED DESCRIPTION:
The aim of this longitudinal study is to investigate whether illness perceptions predict dizziness handicap following a treatment as usual 8-week vestibular rehabilitation programme in patients with chronic vertigo and dizziness.

Participants will be recruited consecutively from patients attending the dizziness and balance exercise programme at Guys & St Thomas' NHS Foundation Trust. Consenting patients will complete the following questionnaires before and after rehabilitation:

1. The Dizziness Handicap Inventory (DHI)
2. The Illness Perceptions Questionnaire - Revised (IPQ-R)
3. The Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS)

The Dizziness Handicap Inventory (DHI) at discharge will be the dependent variable. We will also demographic data including age, gender, and illness type.

ELIGIBILITY:
Inclusion Criteria:

* are aged above 18 years old and are enrolled onto the vestibular rehabilitation programme due to chronic dizziness

Exclusion Criteria:

* Patients will be excluded if they have evidence of central nervous system disorders or cannot speak English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with dizziness and balance disorders.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory (DHI) | At discharge (final session of physiotherapy), an average of 10 weeks
  DHI at discharge (controlling for baseline DHI in the final analysis). The DHI measures the perceived physically, functionally, and emotionally handicapping effects of dizziness although the total score will be used in this study. It consists of 25 questions, for example "Does walking down the aisle of a supermarket increase your problem?", and participants rate either 'Yes', 'No', or 'Sometimes'. The maximum score is 100 and higher scores represent higher levels of disability and activity restriction.

CONTACTS AND LOCATIONS:
Overall Officials: David Herdman, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's & St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided